CLINICAL TRIAL: NCT02240446
Title: Non-Invasive Brain Stimulation for Clinical Intervention for Medication-Resistant Auditory Hallucinations in Schizophrenia Patients
Brief Title: Non-Invasive Brain Stimulation for Medication-Resistant Auditory Hallucinations in Schizophrenia Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Will no longer be conducted. We have started a different project.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1406M51762; IEM (Other: University of Minnesota)
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Auditory Hallucinations; Schizophrenia
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Experimental): Active tDCS
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator): Sham tDCS
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — 2mA stimulation for 20 minutes twice a day for five consecutive days
  Arms: Active tDCS
Device: Sham tDCS — 2mA for 30 seconds twice a day for five consecutive days
  Arms: Sham tDCS

SUMMARY:
The overarching goal of this project is to expand the traditional expertise in non-invasive neuromodulation at the University of Minnesota towards developing novel neuromodulation approaches using transcranial direct current stimulation (tDCS) for treating schizophrenia patients with medication-resistant auditory hallucinations. The investigators will use tDCS to stimulate prefrontal cortex. TDCS is a non-invasive brain stimulation technique that can modulate brain connectivity. Non-invasive brain neuromodulation will be combined (paired-neuromodulation) with training of a task that requires top-down control of auditory processes. Paired-neuromodulation can potentially be used as a therapeutic intervention to decrease auditory hallucinations in schizophrenia.

DETAILED DESCRIPTION:
25% of schizophrenia (SZ) patients report chronic auditory hallucinations (AH) despite being on medication. Previous research proposed that hyperactivity of the left temporo-parietal cortex (11) and hypoactivity in left dorsolateral prefrontal cortex (DLPFC) (12) are associated with the onset of AH. While temporal cortex hyperactivity has been extensively manipulated with neuromodulation interventions trying to reduce AH, results have not been consistent (1,13). Recent transcranial direct current stimulation (tDCS) work that targeted both regions above by applying excitatory stimulation over the left DLPFC and inhibitory stimulation on the left temporo-parietal cortex reported a 30% reduction in AH in patients with medication refractory AH that lasted up to 3 months after treatment (14). The investigators are interested to further investigate whether the use of paired neuromodulation (P-NM) with tDCS in co-targeting top-down executive control with bottom-up sensory processes would result in a larger reduction in AH. To date, there are no studies that have used P-NM to examine the magnitude of plasticity of executive control on sensory processing in SZ patients. This type of P-NM would be relevant since AH are thought to be the result of a lack of top-down control over perceptual distortions of internally generated speech. In the forced-attention dichotic listening task (DL), two different syllables are simultaneously presented to the left and the right ear. Subjects are required to pay attention to and report either the left or right ear stimulus. Due to the preponderance of the contralateral pathways, the right ear syllable is projected to the left temporal lobe for processing, while the left ear stimulus is projected to the right temporal lobe and has to be transferred across the corpus callosum to be processed in the left hemisphere. Healthy controls show a right ear advantage (REA) while SZ patients do not (15). DL task performance requires top-down control over auditory cortex and has been associated with increased DLPFC activation in controls (16). Worse performance in this task has been associated with greater severity of AH (17).

SPECIFIC AIMS: The overall aim is to examine the efficacy of tDCS intervention combined with sensory gating training (paired neuro-modulation; P-NM) to reduce hallucinations (as measured by Positive and Negative Syndrome Scale and the Auditory Hallucination Rating Scale). The investigators will collect pilot data to explore the magnitude of DLPFC plasticity during executive control on auditory processing using P-NM and its effect on hallucination-related behavior. The investigators will combine tDCS to enhance left DLPFC activity with auditory stimuli presented to the right ear. The investigators will use the DL task to assess plasticity of top-down control over auditory sensory perception before and after intervention. The investigators will correlate DL task performance to the magnitude of left DLPFC plasticity and with AH severity.

The investigators hypothesize that (a) DLPFC enhancement will facilitate REA in SZ patients by supporting inhibition of attention to irrelevant syllable and facilitating attention to the right ear syllable; (b) continued pairing of left DLPFC activity and auditory processing will reduce auditory hallucinations (as measured by Positive and Negative Syndrome Scale and the Auditory Hallucination Rating Scale).

Methods: The investigators will recruit 50 SZ patients with persistent severe AH despite medication as measured by the Positive and Negative Syndrome Scale and the Auditory Hallucination Rating Scale (AHRS). To examine the effects of P-NM over time, patients will receive transcranial direct current stimulation (tDCS) during five days, twice a day while they practice the dichotic listening task (DL; Hugdahl 2013). During the DL task, patients will be presented with consonant-vowel syllables via headphones. The syllables will consist of paired presentations of the six stop-consonants /b/, /d/, /g/, /p/, /t/, and /k/ together with the vowel /a/ to form dichotic consonant-vowel syllable pairs of the type /ba - ga/,/ta - ka/ etc. The syllables were paired with each other for all possible combinations, thus yielding 36 dichotic pairs, including the homonymic pairs. Patients will be given two different instructions. In one instruction condition they will be told to focus attention to and report from the right ear, and if think they hear something in the left ear, this should be ignored ("forced-right" condition). In the other condition, patients will be asked to focus attention to and report from the left ear, and if they think that they hear something in the right ear, this should be ignored ("forced-left" condition).

Participants will receive either active tDCS treatment or sham stimulation while performing the DL task. Half of them (n=25) will receive either (a) electrical stimulation (2mA) for 20 minutes to the left DLPFC to enhance top-down control and improve the tuning or gating of the extraneous information or (b) while the other half will receive sham stimulation to control for placebo effects. Active tDCS and sham tDCS will be performed with the same tDCS equipment. The difference is that while active tDCS will be configured to reach constant 2mA stimulation for 20 minutes, sham tDCS will be a very brief 2mA stimulation for 30 seconds. During sham tDCS the subject believes he/she is being stimulated normally, but there should not be any real effects. This same procedure will be repeated during five days, twice a day. At the end of day 5 all patients will complete the Positive and Negative Syndrome Scale and the AHRS to evaluate change in AH. Patients will be asked to complete these scales 3, 6, and 9 months after tDCS intervention to examine long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-V-defined diagnosis of SZ or Schizoaffective Disorder as assessed by the Structured Clinical Interview for Axis I DSM-V Disorders (SCID-I/P)
* Ages 18-45
* Competent and willing to sign consent form

Exclusion Criteria:

* Any serious neurological or endocrine disorder or any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness of more than 30 min, HIV)
* Diagnostic and Statistics Manual (DSM-V) criteria for mental retardation or axis I psychiatric disorder, subjects may have a lifetime but not current diagnosis of depression
* Primary current substance use disorder diagnosis on any substance except for caffeine or nicotine - nicotine use will be recorded but will not be an exclusion criterion
* Medical condition which requires treatment with a medication with psychotropic effects
* Significant risk of suicidal or homicidal behavior
* Documented loss of consciousness (LOC) for longer than 30 minutes or LOC with neurological sequelae
* History of electro-convulsive therapy
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | pre-intervention, post-intervention (after five consecutive days of tDCS intervention), 3,6, and 9 months after post-intervention
  Scores from this scale will show severity of auditory hallucinations. We will assess CHANGE in scores between each time-point described in the Time Frame.

SECONDARY OUTCOMES:
Auditory Hallucination Rating Scale | pre-intervention, post-intervention (after five consecutive days of tDCS intervention), 3, 6, and 9 months after post-intervention
  Depicts severity of auditory hallucination. We will assess CHANGE in scores between each time-point described in the Time Frame.

OTHER OUTCOMES:
Dichotic listening task performance | Will be assessed twice a day for five consecutive days
  Performance measures: Accuracy and reaction time. We will assess CHANGE in task performance between each time-point described in the Time Frame.

CONTACTS AND LOCATIONS:
Overall Officials: Jazmin Camchong, PhD, Principal Investigator — University of Minnesota; Kelvin O Lim, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Background] Hugdahl K, Nygard M, Falkenberg LE, Kompus K, Westerhausen R, Kroken R, Johnsen E, Loberg EM. Failure of attention focus and cognitive control in schizophrenia patients with auditory verbal hallucinations: evidence from dichotic listening. Schizophr Res. 2013 Jul;147(2-3):301-9. doi: 10.1016/j.schres.2013.04.005. Epub 2013 May 9. PMID 23664588
- [Background] Lawrie SM, Buechel C, Whalley HC, Frith CD, Friston KJ, Johnstone EC. Reduced frontotemporal functional connectivity in schizophrenia associated with auditory hallucinations. Biol Psychiatry. 2002 Jun 15;51(12):1008-11. doi: 10.1016/s0006-3223(02)01316-1. PMID 12062886
- [Background] Thomsen T, Rimol LM, Ersland L, Hugdahl K. Dichotic listening reveals functional specificity in prefrontal cortex: an fMRI study. Neuroimage. 2004 Jan;21(1):211-8. doi: 10.1016/j.neuroimage.2003.08.039. PMID 14741658